CLINICAL TRIAL: NCT00834587
Title: A Relative Bioavailability Study of 5 mg Glipizide/500 mg Metformin Hydrochloride Tablets Under Non-Fasting Conditions.
Brief Title: 5 mg Glipizide/500 mg Metformin Hydrochloride Tablets, Non-Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R04-0477
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — metaglip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glipizide Metformin (Experimental): Glipizide Metformin Hydrochloride 5/500 mg Tablet (test) dosed in first period followed by Metaglip™ 5/500 mg Tablet (reference) dosed in second period
  Interventions: Drug: 5 mg/500 mg Glipizide Metformin Hydrochloride Tablets
- Metaglip™ (Active Comparator): Metaglip™ 5/500 mg Tablet (reference) dosed in first period followed by Glipizide Metformin Hydrochloride 5/500 mg Tablet (test) dosed in second period
  Interventions: Drug: 5 mg/500 mg METAGLIP™ Tablets

INTERVENTIONS:
Drug: 5 mg/500 mg METAGLIP™ Tablets — 1 x 5 mg/500 mg, single-dose non-fasting
  Arms: Metaglip™
Drug: 5 mg/500 mg Glipizide Metformin Hydrochloride Tablets — 1 x 5 mg/500 mg, single-dose non-fasting
  Arms: Glipizide Metformin

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 5 mg Glipizide/500 mg Metformin Hydrochloride Tablets manufactured by TEVA Pharmaceutical Industries, Ltd., and distributed by TEVA Pharmaceuticals USA with that of 5 mg/500 mg METAGLIP™ Tablets by Bristol-Myers Squibb Company following a single oral dose (1 x 5 mg/500 mg tablet) in healthy adult subjects administered under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All subjects selected for this study will be healthy men and women 18-45 years of age, inclusive, at the time of dosing. The subject's body mass index (BMI) should be less than or equal to 30.
* Screening Procedures: Each subject will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.

Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.

The screening clinical laboratory procedures will include:

* Hematology: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count;
* Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase; HIV antibody, hepatitis B surface antigen, and hepatitis C antibody screens;
* Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
* Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates, and phencyclidine.
* Serum Pregnancy Screen

If female and:

* of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condom with spermicide, diaphragm with spermicide, intrauterine device (IUD), or abstinence; or
* is postmenopausal for at least 1 year; or
* is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Subjects with a recent history of drug or alcohol addiction or abuse.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a reactive hepatitis B surface antigen screen, a reactive hepatitis C antibody screen, or a reactive HIV antibody screen.
* Subjects demonstrating a positive drug abuse screen when screened for this study.
* Female subjects demonstrating a positive pregnancy screen.
* Female subjects who are currently breastfeeding.
* Subjects with a history of allergic response(s) to glipizide, metformin hydrochloride, or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Subjects who currently use or report using tobacco products within 90 days of Period I dose administration.
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Subjects who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Subjects who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 28 days prior to Period I dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to Period I dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (2):
- United States (2):
  - PRACS Institute Ltd., East Grand Forks, Minnesota
  - PRACS Institute, Ltd., Fargo, North Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- Glipizide Metformin (Test) First: Glipizide Metformin Hydrochloride 5/500 mg Tablet (test) dosed in first period followed by Metaglip™ 5/500 mg Tablet (reference) dosed in second period
- Metaglip™ (Reference) First: Metaglip™ 5/500 mg Tablet (reference) dosed in first period followed by Glipizide Metformin Hydrochloride 5/500 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Glipizide Metformin (Test) First | Metaglip™ (Reference) First
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Glipizide Metformin (Test) First | Metaglip™ (Reference) First
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Glipizide Metformin (Test) First | Metaglip™ (Reference) First
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glipizide Metformin (Test) First | Metaglip™ (Reference) First | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 8 | 14 | 22
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 17 | 18 | 35
  Asian | 1 | 0 | 1
  Black | 1 | 1 | 2
  Native Anerican | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration) - Glipizide in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Glipizide Metformin: Glipizide Metformin Hydrochloride 5/500 mg Tablet (test) dosed in either period
- Metaglip™: Metaglip™ 5/500 mg Tablet (reference) dosed in either period
Arm/Group | Glipizide Metformin | Metaglip™
Number analyzed (Participants) | 39 | 39
ng/mL | 377.949 (92.6166) | 381.282 (96.1909)
Statistical Analysis 1: Comparison: Glipizide Metformin vs Metaglip™; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 99.1, 90% CI [92.4 to 106.2] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf [Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)] - Glipizide
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glipizide Metformin | Metaglip™
Number analyzed (Participants) | 39 | 39
ng*h/mL | 2214.7 (664.87) | 2204.7 (674.77)
Statistical Analysis 1: Comparison: Glipizide Metformin vs Metaglip™; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 100.7, 90% CI [98.8 to 102.6] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t [Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)] - Glipizide
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glipizide Metformin | Metaglip™
Number analyzed (Participants) | 39 | 39
ng*h/mL | 2197.6 (659.57) | 2188.2 (668.99)
Statistical Analysis 1: Comparison: Glipizide Metformin vs Metaglip™; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 100.6, 90% CI [98.8 to 102.5] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

4. Primary Outcome: Cmax (Maximum Observed Concentration) - Metformin in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Glipizide Metformin | Metaglip™
Number analyzed (Participants) | 39 | 39
ng/mL | 661.03 (149.301) | 644.64 (111.631)
Statistical Analysis 1: Comparison: Glipizide Metformin vs Metaglip™; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 101.7, 90% CI [97.3 to 106.3] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

5. Primary Outcome: AUC0-inf [Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)] - Metformin
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis. Data from one completed subject could not be used to estimate AUC0-inf.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glipizide Metformin | Metaglip™
Number analyzed (Participants) | 39 | 38
ng*h/mL | 4397.8 (911.72) | 4423.2 (781.62)
Statistical Analysis 1: Comparison: Glipizide Metformin vs Metaglip™; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 99.2, 90% CI [96.5 to 102.0] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

6. Primary Outcome: AUC0-t [Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant) - Metformin
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glipizide Metformin | Metaglip™
Number analyzed (Participants) | 39 | 39
ng*h/mL | 4220.7 (900.20) | 4233.5 (750.65)
Statistical Analysis 1: Comparison: Glipizide Metformin vs Metaglip™; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 99.1, 90% CI [96.5 to 101.8] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.